CLINICAL TRIAL: NCT03969316
Title: The Comparison of Ultrasound-Guided Transversus Abdominis Plane Block and Quadratus Lumborum Block in The Pediatric Population Undergoing Orchiopexy. A Randomized Controlled Trial
Brief Title: Transversus Abdominis Plane Block Versus Quadratus Lumborum Block in The Pediatric Population Undergoing Orchiopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ozgecan Piril Zanbak, Resident Medical Doctor, Anesthesiology and Reanimation Department, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 71381
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Pain, Postoperative
Keywords: quadratus lumborum block; transversus abdominis plane block; pediatric patient; orchiopexy; regional anesthesia; pain
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block (Active Comparator): After the premedication with ketamine and midazolam will be performed, the patient will be brought to the operation room. After the induction with thiopental 5mg/kg, fentanyl 1mcg/kg, rocuronium 0.6mg/kg, patients will be intubated. The maintenance of the anesthesia will be provided with sevoflurane. 0.4 ml/kg %0.25 bupivacaine will be used as a local anesthetic agent in both groups and the local anesthetic agent will be administrated with ultrasound at the anterolateral border of quadratus lumborum muscle with 18, 20 or 22 Gauge IV Cannula (Bicakcilar Cooperation, Istanbul, Turkey) according to age and body weight.
  Interventions: Procedure: Transversus abdominis plane block, Quadratus lumborum block
- Transversus Abdominis Plane Block (Active Comparator): After the premedication with ketamine and midazolam will be performed, the patient will be brought to the operation room. After the induction with thiopental 5mg/kg, fentanyl 1mcg/kg, rocuronium 0.6mg/kg, patients will be intubated. The maintenance of the anesthesia will be provided with sevoflurane. 0.4 ml/kg %0.25 bupivacaine will be used as a local anesthetic agent in both groups and the local anesthetic agent will be administrated with ultrasound between internal oblique and transversus abdominis muscle with 18, 20 or 22 Gauge IV Cannula (Bicakcilar Cooperation, Istanbul, Turkey) according to age and body weight.
  Interventions: Procedure: Transversus abdominis plane block, Quadratus lumborum block

INTERVENTIONS:
Procedure: Transversus abdominis plane block, Quadratus lumborum block — The TAP block which is one of the abdominal truncal blocks is performed with the blockage of the nerve group which innervates the anterior abdominal muscle wall layers. However, in QL block, the local anesthetic agent spreads through the abdominal wall and paravertebral space with the help of the perimuscular fascia to maintain the somatic analgesia.

SUMMARY:
Transversus abdominis plane (TAP) and Quadratus lumborum (QL) blocks are used for the management of acute pain treatment, especially after the lower and upper abdominal surgeries.

The TAP block which is one of the abdominal truncal blocks is performed with the blockage of the nerve group which innervates the anterior abdominal muscle wall layers. However, in QL block, the local anesthetic agent spreads through the abdominal wall and paravertebral space with the help of the perimuscular fascia to maintain the somatic analgesia.

The investigators' aim in this study, to investigate the effect of the TAP and QL blocks on peroperative and postoperative analgesic consumption in children undergoing unilateral elective orchiopexy.

DETAILED DESCRIPTION:
American Society of Anesthesiologists Physical Status Classification System (ASA) class I-III, aged 6 month-12 years old children undergoing unilateral elective orchiopexy with general anesthesia will be recruited, after the informed consent will be obtained from the parents of the patients, in this randomized controlled trial.

After the premedication with ketamine and midazolam will be performed, the patient will be brought to the operation room. After the induction with thiopental 5mg/kg, fentanyl 1mcg/kg, rocuronium 0.6mg/kg, patients will be intubated. The maintenance of the anesthesia will be provided with sevoflurane.

Subsequently, before the surgery, the patients will be randomized and separated into 2 groups. The investigators will apply the QL block to the first group and TAP block to the other group. 0.4 ml/kg %0.25 bupivacaine will be used as a local anesthetic agent in both group.

In the peroperative period, if the additional analgesia will necessary, remifentanyl 0.1mcg/kg/min will be started, and dosage will be adjusted according to heart rate and blood pressure. If the blood pressure or heart rate will increase more than 20% from the preoperative basal value will be defined as the need for the analgesia.

In the postoperative period, all cohort will be assessed by a blinded investigator at the 10,20,30th minutes, 1,2nd hours in the recovery room, 6th hour in the surgical ward, Face, Legs, Activity, Cry, Consolability Scale (FLACC) will be used for the pain evaluation. 16th and 24th hours will be monitored by the telephone visit from the parents, the pain will be evaluated with the Wong-Baker Faces Pain Rating Scale due to the same-day surgery concept.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* Undergoing elective unilateral orchiopexy

Exclusion Criteria:

* Not giving a consent
* ASA physical status IV
* Need to postoperative ICU care
* History of allergic reactions to anesthetics
* Infection at the injection site
* Laparoscopic Orchiopexy

Ages: 6 Months to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Total Analgesia Consumption | 24 hour
  The required analgesic consumption within the framework of the predetermined protocol will be recorded by the nurses and doctors who do not know which block is used. After discharge, the family will be called by phone to find out the amount of additional analgesic need.
The Effect on Perioperative and Postoperative Pain | 24 hour
  The investigator will screen and record perioperative hemodynamic parameters for the perioperative pain evaluation. The Face, Legs, Activity, Cry, Consobility (FLACC) Score will be used for evaluation of the postoperative pain. The FLACC pain assessment score is evaluated out of 10 points. While a score of zero defined as no pain, 1-3 is mild pain, 4-6 is moderate pain, 7-10 is severe pain, respectively. If the score is 4 and above, additional analgesic administration will be planned.
The Effect on Post-discharge Pain | 24 hour
  Post-discharge pain will be assessed by the Wong Baker Score. Pain will be evaluated based on six facial expressions between zero and ten points. If the score is four or more, additional analgesic administration will be planned.

SECONDARY OUTCOMES:
Parent satisfaction score | 24 hour
  At the postoperative 24th hour, the investigator will ask to the parents by telephone visit. Parent satisfaction score is defined as unsatisfied (1), partially satisfied (2), satisfied (3)

CONTACTS AND LOCATIONS:
Overall Officials: Ozgecan P Zanbak, MD, Principal Investigator — Istanbul University - Cerrahpasa; Ayse C Tutuncu, MD,Prof, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488
- [Background] Oksuz G, Bilal B, Gurkan Y, Urfalioglu A, Arslan M, Gisi G, Oksuz H. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Children Undergoing Low Abdominal Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):674-679. doi: 10.1097/AAP.0000000000000645. PMID 28759502
- [Derived] Mutlu OPZ, Tutuncu AC, Kendigelen P, Kara Esen B. Posterior transversus abdominis plane block versus lateral quadratus lumborum block in children undergoing open orchiopexy: a randomized clinical trial☆. Braz J Anesthesiol. 2024 Sep-Oct;74(5):744443. doi: 10.1016/j.bjane.2023.06.004. Epub 2023 Jul 8. PMID 37429376